CLINICAL TRIAL: NCT01634126
Title: Maximizing Yield of the Fecal Immunochemical Test for Colorectal Cancer Screening
Acronym: MY-FIT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 5R01CA154982 (NIH); 1R01CA154982 (NIH)
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: Colon; Rectal; Cancer; Screening; FIT; Fecal
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 FIT kit (Active Comparator)
  Interventions: Behavioral: 1 FIT kit
- 2 FIT kit (Active Comparator)
  Interventions: Behavioral: 2 FIT kit

INTERVENTIONS:
Behavioral: 1 FIT kit — Patient receives 1 FIT
  Arms: 1 FIT kit
Behavioral: 2 FIT kit — Patient receives 2 FIT kits
  Arms: 2 FIT kit

SUMMARY:
Colorectal cancer (CRC) is a leading cause of cancer death in the United States. Screening for CRC reduces CRC mortality, yet rates of screening in the United States remain low. Fecal occult blood testing (FOBT) has an established positive balance of benefit and risk, is the least expensive, and is the preferred method for nearly half of patients. A newer fecal screening test, the fecal immunochemical test (FIT), offers significant improvements over the FOBT. It is easier to use and is more sensitive at detecting both CRC and precancerous adenomas than the FOBT. The OC-Micro FIT is of particular interest because it is highly sensitive and specific and it is the only FIT test approved in the US that can be processed in an automated manner. Thus, the OC-Micro is an optimal method for use in mass screening programs to improve community CRC-screening rates. However, prior studies of OC-Micro suffer from several limitations: they were conducted in populations not optimal for assessing screening performance in average risk patients in the U.S. and the studies did not clearly establish optimal number of samples required and cut-points for test positivity. Therefore, the overall goal of MY-FIT is to capitalize on the highly integrated and extensive electronic medical record system of the study site to collect two separate sets of data that, when synthesized, will provide a thorough picture of the comparative patient adherence to, sensitivity, specificity, and costs of different protocols for using the OC-Micro FIT. Specifically, among KPNW members aged 50-75 who are at average risk for colorectal cancer (CRC) and who are due for CRC screening (n=78,000), the investigators propose to:

1. Compare the sensitivity, specificity, positive predictive value, and negative predictive value for colorectal cancer and advanced adenoma (advanced neoplasia) between a single-sample FIT (1-FIT) and a two-sample FIT (2-FIT) using varying cut points for a positive test (n=2100).
2. Compare patient adherence to completion of a 1-FIT versus a 2-FIT protocol (n=3000).
3. Assess and compare cost per screen for a 1-FIT versus a 2-FIT protocol, and the cost per advanced neoplasia detected in a 1-FIT versus a 2-FIT protocol (using varying cut points for a positive test) (n=78,000).

Answering the above questions will provide a much-needed strong evidence base for a best-practice, cost-effective method of using the OC-Micro FIT to screen for CRC in a general U.S. population.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for standard KPNW automated telephonic colorectal cancer screening reminder and have indicated on the call that they wish to screen with FIT.

Exclusion Criteria:

* Kaiser Permanente members less than 1 year.
* Currently on the Kaiser Permanente Center for Health Research Do Not Call list.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2761 (Actual)
Dates: Start 2012-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
FIT Kit adherence | Year 2 of study
  Among KPNW members aged 50-75 who are at average risk for colorectal cancer (CRC) and who are due for CRC screening, we propose to compare patient adherence to completion of a 1-FIT versus a 1-2 FIT protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Liles, MD, Principal Investigator — Kaiser Foundation Hospital
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States